CLINICAL TRIAL: NCT04970277
Title: Efficacy of Drinking Water on Transit Time and Complete Examination Rate During Capsule Endoscopy
Brief Title: Efficacy of Drinking Water During Capsule Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, doctoral supervisor of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021SDU-QILU-054
Record Dates: First submitted 2021-07-18; First posted 2021-07-21 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Capsule Endoscopy
Keywords: Capsule endoscopy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drinking water group (Experimental): Patients in this group drink colorless water after capsule ingestion.
  Interventions: Other: drinking water group
- control group (Other): Patients in this group don't drink colorless water after capsule ingestion.
  Interventions: Other: control group

INTERVENTIONS:
Other: drinking water group — Those randomized to drink water group were asked to drink 200 mL colorless water every 10 minutes, starting at the time of capsule ingestion until three times in total.
  Arms: drinking water group
Other: control group — Those randomized to control group were asked not to drink extra water after capsule ingestion.
  Arms: control group

SUMMARY:
The aims of this study are to evaluate the effect of early drinking water after the capsule ingestion on the gastrointestinal transit and image quality of capsule endoscopy.

DETAILED DESCRIPTION:
Capsule endoscopy has been a significant technologic advancement that has allowed the direct examination of mucosa throughout the entire small intestine in a noninvasive fashion; and it has become the primary technique for imaging the small bowel. However, as imaging time is limited to about 8 hours, a prolonged transit of the capsule endoscope in the stomach may result in an incomplete small bowel transit (i.e. failure of the capsule to reach the cecum). Delayed transit time of stomach may be responsible for the failure of capsule endoscopy to visualize the distal portions of the small bowel, and potentially may result in the inability to identify small-bowel pathology in these areas. Previous study showed that drinking water might improve completion rate of capsule endoscopy. And bowel preparation of clear liquids may improve image quality of small bowel mucosa. The aim of this study was to assess the effect of drinking water on the transit time，completion rate and image quality of capsule endoscopy.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-80 years undergoing capsule endoscopy

Exclusion Criteria:

1. Patients with suspected intestinal obstruction, intestinal diverticulum, stricture or fistula
2. previous gastric or small-bowel surgery
3. pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-07-18 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
gastric transit time | 3 months
  the time between the first gastric image and the first duodenal image
small-bowel transit time | 3 months
  the imaging time of capsule endoscopy in the small bowel

SECONDARY OUTCOMES:
complete examination rate of the small bowel | 3 months
  the percentage of patients with complete examination of the small bowel in each group
image quality | 3 months
  The scale was based on the uncovered image area percentage (0, 0%-20%; 1, 20%-40%; 3, 60%-80%; 4, 80%-100%). The image quality was based on the mean of 5-min scores and higher scores mean a better outcome.
diagnostic yields | 3 months
  Clinical diagnoses made by the capsule endoscopy were recorded for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD, PhD, Principal Investigator — Shandong University Qilu hosipital, China
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China